CLINICAL TRIAL: NCT02239939
Title: Weighted Vest Use to Preserve Muscle and Bone During Obesity Treatment for Osteoarthritis
Brief Title: Arthritis Pilot for Preserving Muscle While Losing Weight
Acronym: APPLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Medifast, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00028928
Record Dates: First submitted 2014-09-09; First posted 2014-09-15 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Obesity; Osteoarthritis
Keywords: older adults, body composition, weight loss, muscle mass
MeSH Terms: conditions — Obesity; Osteoarthritis; Weight Loss | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vest + Diet (Experimental): All participants will undergo a 22 week dietary weight loss. In addition, participants will be asked to wear a weighted vest for >10 hours a day. Weight in the vest is adjusted to match weight lost during the intervention.
  Interventions: Behavioral: Vest; Behavioral: Diet
- No Vest + Diet (Active Comparator): All participants will undergo a 22 week dietary weight loss intervention. Participants in this group will be asked not to change their daily habits other than adherence to the diet protocol.
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Vest — light weight, adjustable, vest to be worn underneath clothes that weight can be added to
  Other Names: Hyperwear Vest Pro
  Arms: Vest + Diet
Behavioral: Diet — Participants will undergo a 22 week dietary weight loss intervention which will incorporate dietary practices for achieving weight loss while minimizing muscle and bone loss. Participants will be instructed by the Registered Dietitian to follow a low calorie diet. Individual calorie goals will be adjusted during the study if necessary to achieve a targeted weight loss goal of at least 8%, but no more than 12%, within the intervention time frame.
  Other Names: Medifast 4&2&1

SUMMARY:
The purpose of this research study is to see whether wearing a weighted vest during a period of active weight loss can decrease the loss of muscle and bone that occurs during weight loss. We will also determine if study participants who wear the weighted vest will have greater improvements in physical function and self-reported disability, pain, stiffness, fatigue and quality of life. This knowledge could impact weight loss programs designed for older adults.

Hypothesis: Participants randomized to VEST will experience similar weight loss, but less loss of lean mass and bone density, than participants randomized to Control.

DETAILED DESCRIPTION:
The loss of muscle mass and bone density during weight loss is partially attributed to the decrease in mechanical stress on these tissues as weight is reduced. As a result, performing exercises that enhance muscle and gravitational loading during the period of caloric restriction usually diminishes the relative amount of muscle and bone loss for a given weight loss, but these interventions do not fully prevent all muscle and bone loss.In addition, conventional exercise training interventions often require expensive equipment, on-site participation, and, ideally for older, obese adults, safety supervision by trained exercise leaders. Moreover, the exercises performed may not fully translate into improvement in daily tasks due to training specificity, and are not always tolerated or sustained, especially in obese persons with OA. On the other hand, it is conceivable that treating the decrease in mechanical load from weight loss by externally replacing lost weight via use of a weighted vest may also be effective for reducing muscle and bone loss during caloric restriction. In animal models, mechanisms regulating skeletal tissue structure and function respond in a similar fashion to increases in actual or externally-added body mass. Also, research shows that exercising while wearing weighted vests can improve bone density, muscle mass, and lower extremity strength in older adults. However, no prior studies have examined the effects of weighted vest use on muscle mass and bone density during a period of intentional weight loss.

The main objective of this pilot study is to assess feasibility (accrual, retention, compliance) of daily use of a weighted vest during a diet intervention, to estimate the variability of outcome measures, and to obtain preliminary estimates of treatment efficacy. A controlled, randomized design will be used so we can obtain a realistic estimate of accrual and an unbiased estimate of treatment efficacy.

A total of 36 older (age=65-79 yrs), obese (BMI=30-40 kg/m2), sedentary men and women with x-ray evidence of knee OA will undergo a 22 week weight loss intervention (targeting 10% weight loss) with randomization to one of two groups (n=18/grp): 1) No vest use (Control); or 2) Progressive weighted vest use during normal daily activities (VEST).

ELIGIBILITY:
Inclusion Criteria:

* BMI=30-40 kg/m2; Wt<135 kg,
* self- reported MD diagnosis of osteoarthritis
* No evidence of clinical depression or other contraindications for participation in voluntary weight loss,
* Sedentary lifestyle (<30 min, 3 d/wk of exercise),
* Able to provide own transportation to study visits and intervention,
* Not dependent on a cane or walker,
* Willing and able to consume meal replacement products,
* Not involved in other research study,
* Approved for participation by Medical Director,
* Willing to provide informed consent.

Exclusion Criteria:

* Weight loss or gain (±5%) in past 6 mos,
* Excessive alcohol use (> 14 drinks/wk),
* Smoker (>1 cigarette/d or 4/wk within yr),
* Evidence of cognitive impairment (MoCA score <22) or difficulty with hearing or vision that would interfere with study participation, Insulin-dependent or uncontrolled diabetes (FBG >125 mg/dl) or Hypertriglyceridemia (TG>400 mg/dl),
* Osteoporosis (T-score< -2.5 on hip or spine); Hip fracture, joint replacement, or spinal surgery in past 6 mos, or hyperkyphosis,
* Uncontrolled hypertension (BP>160/90 mmHg) or abnormal kidney or liver tests per Medical Director discretion,
* Self- reported hepatitis B or C,
* Severe anemia (Hb<10 g/100 ml),
* Past or current uncontrolled endocrine/metabolic disease, neurological or hematological disease, fibromyalgia, chronic pulmonary disease, hyperparathyroidism, rheumatoid arthritis, unstable angina, MI, cardiac surgery within 3 months,
* Cancer requiring treatment in past year except non-melanoma skin cancers,
* Regular use of medications that may influence body weight, hormones, weight loss medications, bone remodeling medication, prior use of medications that affect bone, insulin-dependent,
* Unable to tolerate vest run-in.

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Nicklas, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health Sticht Center on Aging, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available upon email request to the study PI and upon completion of a data-sharing agreement. This agreement will require that data be used only for research purposes, that no attempts be made to identify individual patients, that the data will be kept secure, that the user will not distribute the data to other researchers, that the user will return the files or destroy them once the project is completed, and that the user will acknowledge the data source. All data files will be de-identified. In addition, variables that could permit linkages to individual research participants and variables that could lead to deductive disclosure of the identity of individual subjects will be removed or recoded. We will create a link on our website that describes our study and the data available for data sharing with descriptions.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vest + Diet | No Vest + Diet
Started | 20 | 17
Completed | 18 | 15
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vest + Diet | No Vest + Diet | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (3.4) | 69.9 (2.6) | 70.1 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 17 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 16 | 12 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Lean Mass Measured by DXA
Description: Lean body mass (Whole body and lower-extremity lean mass are used in total calculation).
Time Frame: Baseline and 22 weeks
Measure: Mean (Standard Deviation); unit: Kg
Groups:
- Diet+Vest: All participants will undergo a 22 week dietary weight loss. In addition, participants will be asked to wear a weighted vest for >10 hours a day. Weight in the vest is adjusted to match weight lost during the intervention.
  Vest: light weight, adjustable, vest to be worn underneath clothes that weight can be added to
  Diet: Participants will undergo a 22 week dietary weight loss intervention which will incorporate dietary practices for achieving weight loss while minimizing muscle and bone loss. Participants will be instructed by the Registered Dietitian to follow a low calorie diet. Individual calorie goals will be adjusted during the study if necessary to achieve a targeted weight loss goal of at least 8%, but no more than 12%, within the intervention time frame.
- No Vest+Diet: All participants will undergo a 22 week dietary weight loss.
  Diet: Participants will undergo a 22 week dietary weight loss intervention which will incorporate dietary practices for achieving weight loss while minimizing muscle and bone loss. Participants will be instructed by the Registered Dietitian to follow a low calorie diet. Individual calorie goals will be adjusted during the study if necessary to achieve a targeted weight loss goal of at least 8%, but no more than 12%, within the intervention time frame.
Arm/Group | Diet+Vest | No Vest+Diet
Number analyzed (Participants) | 18 | 15
Kg | -2.9 (1.6) | -2.3 (1.9)

2. Secondary Outcome: Change in Hip Bone Density
Description: Hip bone density as measured by DXA.
Time Frame: Basleine and 22 weeks
Measure: Mean (95% Confidence Interval); unit: g/cm2
Arm/Group | Vest + Diet | No Vest + Diet
Number analyzed (Participants) | 18 | 15
g/cm2 | -6.1 [-15.7 to 3.5] | -18.7 [-29.3 to -8.1]

3. Secondary Outcome: Changes in Self-report on Fatigue Using Pittsburgh Fatigability Scale (PFS)
Description: Pittsburgh Fatigability Scale (PFS) is a self-administered 10 item assessment. It asks participants to rate the level of physical and mental fatigue they experience or imagine after completing a set of hypothetical activities related to daily life at a fixed intensity and duration. The participant provides a score from 0-5 where "0' equals no fatigue at all, and "5" equals extreme fatigue.
Time Frame: baseline and 22 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vest + Diet | No Vest + Diet
Number analyzed (Participants) | 18 | 15
units on a scale | 15.3 (13.6) | 12.3 (14.6)

4. Other Pre Specified Outcome: Change in Body Weight
Description: Body weight
Time Frame: Baseline and 22 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Vest + Diet | No Vest + Diet
Number analyzed (Participants) | 18 | 15
kg | -110.6 (5.7) | -10.9 (4.1)

5. Other Pre Specified Outcome: Changes in Lower Extremity Physical Function
Description: SPPB is a measure of lower-extremity function consisting of walking speed, balance, and repeated chair stands. These 3 performance measures are scored from 0 to 4, with 4 indicating the highest level of performance and 0 the inability to complete the task, with a summary score of 0-12.The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability.
Time Frame: Baseline and 22 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vest + Diet | No Vest + Diet
Number analyzed (Participants) | 18 | 15
units on a scale | 0.1 (0.34) | 0.15 (0.16)

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Vest + Diet | No Vest + Diet
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/20 | 2/17
Other Adverse Events (participants affected / at risk) | 15/20 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vest + Diet (N=20) | No Vest + Diet (N=17)
diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — participant had history of diverticulitis since 1980s until 11/2013 which was cleared by antibiotics. With this episode, participant when to doctor as soon as symptoms started.
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Participant became dehydrated after another illness. participant felt it was due to medications- sudafed and mucinex. Participant was hospitalized overnight.
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Was seen in the Emergency room for bronchitis
chest pain (Cardiac disorders) | 1 (1) | 0 (0) — participant had chest pain. Went to hospital and ended up having a blockage that required a stent
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vest + Diet (N=20) | No Vest + Diet (N=17)
back spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pulled back muscle/ back pain/ neck pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
bronchitis/pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
diarrhea/nausea/stomach virus (Gastrointestinal disorders) | 3 (3) | 0 (0)
Tripped and fell (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
sinus infection/cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
compression fracture in spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
twisted knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
injured by fallen debri (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
fracture in ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
dizzy while standing (Ear and labyrinth disorders) | 0 (0) | 1 (1)
lesion removed from under eye (Eye disorders) | 0 (0) | 1 (1)
vericous vein swelling (Vascular disorders) | 1 (1) | 0 (0)
tingling/numbness in back/arm (Nervous system disorders) | 1 (1) | 0 (0)
drug reaction to sulfamethaxayole (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pulled muscle in shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
oxygen level drops at night (General disorders) | 0 (0) | 1 (1)
lower lip swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
gout flare up (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
spinal column pressing on nerves (Nervous system disorders) | 1 (1) | 0 (0)
pinch in back (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No